CLINICAL TRIAL: NCT00023881
Title: Phase II Study of a Proteasome Inhibitor, PS-341 (NSC 681239) in Chronic Myelogenous Leukemia (CML) in Chronic or Accelerated Phase
Brief Title: Bortezomib in Treating Patients With Chronic Myelogenous Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068872; MDA-DM-00274; NCI-1756; DM00-274 (Other: UT MD Anderson Cancer Center)
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of bortezomib in treating patients who have chronic myelogenous leukemia in chronic or accelerated phase.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of bortezomib, in terms of response rate, duration of response, and survival of patients with Philadelphia chromosome-positive chronic myelogenous leukemia in chronic or accelerated phase.
* Assess the toxicity of this drug in these patients.

OUTLINE: Patients receive bortezomib intravenous (IV) over 3-5 seconds twice weekly on weeks 1-2. Treatment repeats every 3 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 5-30 patients will be accrued for this study within 15-30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Philadelphia (Ph) chromosome-positive chronic myelogenous leukemia (CML) in chronic or accelerated phase, defined as having any of the following:

  * Peripheral blood (PB) or bone marrow (BM) blasts at least 10% but less than 30%
  * PB or BM blasts and promyelocytes at least 20%
  * PB or BM basophils at least 20%
  * Progressive splenomegaly (at least 10 cm confirmed twice at least 4 weeks apart or 50% increase in splenomegaly over 4 weeks)
  * Clonal evolution defined as the presence of additional cytogenetic abnormalities other than the Ph chromosome
  * Thrombocytopenia (platelet count less than 100,000/mm^3) unrelated to therapy
  * Hemoglobin less than 7 g/dL unrelated to therapy or bleeding
* Failed prior treatment with imatinib mesylate or intolerant, unable, or unwilling to receive it
* Ineligible for higher-priority or higher-efficacy regimens or protocols
* No blastic phase CML

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy:

* At least 18 weeks

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Other:

* No other concurrent illness that would preclude study entry
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No more than 2 prior cytotoxic regimens in addition to imatinib mesylate and/or hydroxyurea
* At least 4 weeks since prior chemotherapy and recovered
* Concurrent hydroxyurea and/or anagrelide allowed during first 2 courses

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* See Disease Characteristics
* See Chemotherapy
* At least 24 hours since prior imatinib mesylate
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2001-07-02 (Actual); Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center at University of Texas, Houston, Texas, United States